CLINICAL TRIAL: NCT07222241
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Adjunct Nerve Blocks in Mohs Micrographic Surgery on the Face and Scalp
Brief Title: Comparing Numbing Techniques in Mohs Micrographic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UPCC 10625
Record Dates: First submitted 2025-10-22; First posted 2025-10-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Skin Cancer Face; Skin Cancer Scalp
Keywords: Mohs; Nerve block
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Nerve Block (Placebo Comparator): Placebo regional nerve block with sterile normal saline plus local anesthetic infiltration of the tumor site.
  Interventions: Other: Placebo Nerve Block
- Regional Nerve Block (Experimental): Adjunct regional nerve block with lidocaine plus local anesthetic infiltration of the tumor site.
  Interventions: Other: Nerve Block

INTERVENTIONS:
Other: Nerve Block — 0.45% lidocaine with 1:200,000 epinephrine
  Arms: Regional Nerve Block
Other: Placebo Nerve Block — Sterile normal saline
  Arms: Placebo Nerve Block

SUMMARY:
This study seeks to determine whether adjunct regional nerve blocks reduce pain and anxiety in adult patients undergoing Mohs micrographic surgery for face and scalp skin cancers. Participants will be randomized to one of two arms: (1) placebo regional nerve block with sterile normal saline or (2) adjunct regional nerve block with lidocaine. All patients receive local infiltration with lidocaine for complete anesthesia.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-center clinical trial involving adult patients undergoing Mohs micrographic surgery for cutaneous malignancy on the face and scalp. Patients will be randomized into one of two study arms:

1. Placebo Nerve Block Group: Placebo regional nerve block with sterile normal saline plus standard local infiltration with 0.45% lidocaine with 1:200,000 epinephrine.
2. Experimental Nerve Block Group: Regional nerve block with 0.45% lidocaine with 1:200,000 epinephrine plus standard local infiltration with 0.45% lidocaine with 1:200,000 epinephrine.

Pain scores and other perioperative outcomes will be measured to assess the impact of these anesthetic techniques on patient experience, surgical efficiency, and analgesic efficacy. Pain will be assessed using a validated 0-10 Visual Analog Scale (VAS), where 0 = no pain and 10 = worst pain imaginable. Patients will rate their pain at three time points on a printed VAS scale: (T1) after nerve block, (T2) immediately after completion of local infiltration but before surgical excision, and (T3) at the end of stage 1 of Mohs micrographic surgery. Anxiety will be assessed using a validated 0-10 VAS (0 = no anxiety, 10 = worst anxiety imaginable) at the same three time points (T1, T2, and T3). Anxiety will also be assessed preoperatively (T0). Patients will be instructed on the use of these scales prior to surgery, and outcome assessors blinded to allocation will record responses verbatim at the specified intervals. Subjects will be randomized in a 1:1 ratio to either of the study arms. Randomization will be performed using a computer-generated sequence. Allocation concealment will be maintained through sealed opaque envelopes or electronic assignment by personnel not involved in outcome assessment. The study is double-blind; neither the patient nor the clinical staff assessing outcomes will be aware of the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Scheduled to undergo MMS.
* Lesions on the face or scalp, defined as the region superior to the mandibular margin anteriorly, superior to the external occipital protuberance posteriorly, and superior to the mastoid processes laterally.
* Tumor diameter plus anticipated stage 1 MMS margin ≥2 cm in diameter OR any tumor on the lip, nose, or eyelid.
* Ability to complete patient reported outcome measures in English.

Exclusion Criteria:

* Known allergy or contraindication to lidocaine or epinephrine.
* Chronic opioid use or pre existing pain disorders that may interfere with pain reporting.
* Presence of scar tissue at the anatomic site of local infiltration or nerve block that may alter anesthetic penetration.
* Concurrent multi site Mohs procedure.
* Signs of skin and soft tissue infection at the anatomic site of local infiltration or nerve block.
* Inability to understand or complete pain and satisfaction assessments.
* Pregnant or breastfeeding.
* Use of sedatives or anxiolytics prior to the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Pain | T1: After nerve block; T2: Immediately after completion of local infiltration but before surgical excision; T3: At the end of stage 1 of Mohs micrographic surgery.
  Pain rating reported by the patient using a Visual Analog Scale (0 = no pain; 10 = worst pain imaginable).

SECONDARY OUTCOMES:
Anxiety | T0: Preoperative; T1: After nerve block; T2: Immediately after completion of local infiltration but before surgical excision; T3: At the end of stage 1 of Mohs micrographic surgery.
  Anxiety rating reported by the patient using a Visual Analog Scale (0 = no anxiety; 10 = worst anxiety imaginable). Exploratory sub-endpoints will investigate the relationship between patient anxiety and pain scales.
Needle Sticks | During local infiltration.
  Number of needle sticks needed during local infiltration to achieve complete anesthesia. Does not include punctures used to assess numbness.
Anesthetic Volume | From the administration of the first nerve block to the end of stage 1.
  Sum of all injected volumes (blocks + infiltration + preventative + rescue). Exploratory sub-endpoints will investigate local infiltration-only volume to estimate sparing effect of nerve blocks.
Rescue Anesthesia | Stage 1 of Mohs micrographic surgery.
  Proportion of participants receiving ≥1 rescue infiltration after anesthesia is complete and before stage-1 end. Exploratory sub-endpoint to investigate the number of rescue events during stage 1.
Patient Satisfaction | Assessed at the end of stage 1 of Mohs micrographic surgery.
  Score from a five-point Likert scale assessing patient satisfaction. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Miller, MD, Principal Investigator — Univerisity of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including clinical assessments) that underlie the results reported in this study will be made available to qualified researchers upon reasonable request. Data will be accessible after publication of the main study findings and for up to 5 years thereafter. Requests should be submitted in writing to the Principal Investigator, and access will be granted following review and approval by the University of Pennsylvania IRB and data use agreements as required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the main study findings and for up to 5 years thereafter
Access Criteria: Requests should be submitted in writing to the Principal Investigator, and access will be granted following review and approval by the University of Pennsylvania IRB and data use agreements as required.